CLINICAL TRIAL: NCT00342784
Title: Genetic Analysis of Cases, Controls, and Families With Prostate Cancer
Brief Title: Identification of Prostate Cancer Genes
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905034; 05-HG-N034
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07-30

CONDITIONS: Prostate Cancer
Keywords: Mutation; Cancer Genetics
MeSH Terms: conditions — Prostatic Neoplasms

SUMMARY:
This study will identify genes that predispose men to prostate cancer and affect the rate and type of disease spread, the aggressiveness of the disease, and the long-term outcome. Several studies show there is a genetic component to prostate cancer susceptibility, and that a first-degree relative with prostate cancer increases a man's risk 2- to 3-fold compared to those without a family history. The risk is significantly higher if the relative was diagnosed at younger than 65 years of age, or if three or more first-degree relatives are affected.

The study will try to locate prostate cancer genes in DNA samples using two methods: linkage analysis and association studies. Traditionally, the search for a disease gene begins with linkage analysis, in which the aim is to find the rough location of the gene relative to another DNA sequence, called a "genetic marker," whose position is already known. In genetic association studies, genes from a large number of patients are compared with healthy controls who are matched by age, race, and geographic region.

DNA samples for this study come from patients in the two following studies at the Fred Hutchinson Cancer Research Center, Seattle, Washington:

Family study: Participants are families with prostate cancer who have: 1) three or more first-degree relatives with prostate cancer; 2) three generations with prostrate cancer either through the maternal or paternal side of the family; or 3) two first-degree relatives with prostate cancer diagnosed before age 65 or who were African American.

Population-based study: Participants are patients with prostate cancer and matched healthy control subjects.

The identification of prostate cancer genes important in susceptibility to the disease and its aggressiveness may permit earlier detection and development of more directed and effective treatments based on underlying genetics.

DETAILED DESCRIPTION:
The notion that there are prostate cancer susceptibility genes has since been suggested by case-control, cohort and twin studies. The effect is strongest among first-degree relatives, where the relative risk estimates range from 1.7 to 3.7. Families reporting younger ages at diagnosis and multiple relatives with prostate cancer were demonstrated even higher relative risks. For example, compared to men with no family history, men with three or more first-degree relatives with prostate cancer have almost an 11-fold increased risk. Although the majority of studies focused on Caucasians, similar elevations in risk associated with a family history of disease have been reported for Asian and African Americans. While the majority of the data seems to point towards autosomal dominant genes, evidence for an X-linked or recessive inheritance has also been reported.

During the last decade, others and we have been devoted to the search for hereditary prostate cancer (HPC) loci either by linkage or by association with candidate genes. A generally agreed upon definition of HPC families now exists. These are families in which there is either: 1) prostate cancer in three or more first-degree relatives; 2) prostate cancer in three successive generations; or 3) a cluster of two relatives diagnosed at less than or equal to 55 years.

Armed with these criteria, others and we have collected large data sets of likely hereditary families and undertaken genome wide scans. However, locus heterogeneity issues have made the task difficult. There are clearly many genes that contribute to prostate cancer susceptibility, and many are likely to be weakly penetrant. We have stratified the data derived from our genome scan by a number of likely factors such as age at diagnosis, number of affected men, founder effects aggressiveness of disease, and presence of other cancers in the family to develop more homogeneous datasets. We propose to continue those sorts of studies, as well as focus on cloning genes in regions we and others have identified to date. To test hypotheses that certain variants are associated with prostate cancer susceptibility or progression of disease, will also conduct association studies in a population-based, case control study of middle aged men with prostate cancer. This will allow us to test the putative association of candidate genes and SNPs in prostate cancer susceptibility, aggressivity, and long-term outcomes.

ELIGIBILITY:
* INCLUSION CRITERIA:

Study families were required to meet at least one of the following criteria:

Have three or more first-degree relatives with PC

Have three generations with PC, either through paternal or maternal lineage; or

Have two-first degree relatives with PC diagnosed before age 65 or who were African American. All surviving men, and selected unaffected men and females were invited to join.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5118 (Actual)
Dates: Start 2004-11-08; Study Completion 2018-07-30

CONTACTS AND LOCATIONS:
Overall Officials: Elaine A Ostrander, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Fincham SM, Hill GB, Hanson J, Wijayasinghe C. Epidemiology of prostatic cancer: a case-control study. Prostate. 1990;17(3):189-206. doi: 10.1002/pros.2990170303. PMID 2235728
- [Background] Steinberg GD, Carter BS, Beaty TH, Childs B, Walsh PC. Family history and the risk of prostate cancer. Prostate. 1990;17(4):337-47. doi: 10.1002/pros.2990170409. PMID 2251225
- [Background] Hayes RB, Liff JM, Pottern LM, Greenberg RS, Schoenberg JB, Schwartz AG, Swanson GM, Silverman DT, Brown LM, Hoover RN, et al. Prostate cancer risk in U.S. blacks and whites with a family history of cancer. Int J Cancer. 1995 Jan 27;60(3):361-4. doi: 10.1002/ijc.2910600315. PMID 7829245